CLINICAL TRIAL: NCT02494011
Title: Closed Kinetic Chain Exercise Versus Russian Current Stimulation in Rehabilitation of Colles' Fracture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, emad eldin mohamed, MD, Closed kinetic chain exercise versus Russian current stimulation in rehabilitation of colles' fracture., October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00300
Record Dates: First submitted 2015-07-04; First posted 2015-07-10 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Distal Radius Fracture
Keywords: Colles' Fracture; CKCE; Russian current
MeSH Terms: conditions — Wrist Fractures; Colles' Fracture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- traditional exercise (group I) (Experimental): Mobilization:2 strokes per one second and repeated 6 times during session
  * stretching exercise: 15 to 20 minutes
  * passive range of motion: 5 minutes at beginning and at end
  * active range of motion: 20 repetition
  * oedema control: 15s active contraction of fingers of 15s relax for 3 times
  Interventions: Other: traditional exercise
- russian current stimulation (group II) (Experimental): The frequency was 2.5 kHz for 15 minutes
  Interventions: Other: traditional exercise; Other: Russian current stimulation
- CKC (group III) (Experimental): wall press exercise - plyometric exercise-Quadruped rhythmic stabilization- press up exercise
  closed kinetic chain exercises performed 10 times and each week 2 more repetitions added as a progression
  Interventions: Other: traditional exercise; Other: closed kinetic chain exercise

INTERVENTIONS:
Other: traditional exercise — mobilization stretching exercise
  Other Names: I
Other: Russian current stimulation — stimulation to wrist flexors for 15 minutes
  Other Names: II
  Arms: russian current stimulation (group II)
Other: closed kinetic chain exercise — wall press exercise plyometric exercise
  Other Names: III
  Arms: CKC (group III)

SUMMARY:
This study compared the effects of closed kinetic chain exercise and Russian current stimulation on pain, functional disability, wrist range of motion (ROM) and grip strength in patients with colles' fracture. Forty five patients with stable colles' fractures are randomly classified into three groups with fifteen patients in each group; Group I received traditional exercise in the form of; Mobilization, stretching exercises, range of motion exercises (passive and active) and edema control of the wrist joint. Group II stimulated by electrical Russian current in addition to traditional exercise. Group III received closed kinetic chain exercise (wall press, plyometric wall push up, Quadruped rhythmic stabilization, and Push up exercises) plus traditional exercise. All outcome measures including Pain, function, Wrist ROM, and grip strength were evaluated before and after the treatment program.

DETAILED DESCRIPTION:
Material and Methods Patients Forty five patients with stable colles' fractures collected from October 6 hospital and elsahel hospital and treated conservatively with closed reduction and casting and after removal of plaster cast they involved in the study from January 2013 to May 2013. All patients were assigned randomly into three groups by drawing of lots; group I (traditional exercise), group II (Russian stimulation) and group III (CKC).

Exclusion criteria were:

1. Patient less than 20 years old.
2. Intraarticular fracture of involved hand.
3. Any problem affects shoulder /elbow joints of the involved side.
4. Nerve lesions.
5. Fracture of ulna.

Intervention

Group I received traditional exercise program in the form of;

1. Mobilization: With patient sitting on high back support chair, gentle traction with oscillatory technique (gliding) for thirty seconds were used to increase wrist range of motion in all directions with the frequency of two strokes per one second and repeated six times during session. For progression ten seconds was added to the frequency of mobilization technique each session.
2. Stretching exercises: Wrist flexors (flexor carpi radialis and flexor carpi ulnaris), extensors (extensor carpi radialis longus and brevis and extensor carpi ulnaris), radial deviators and ulnar deviators were stretched gently within the limit of pain with fifteen to twenty seconds hold at end of creeping movement of contractile and noncontractile elements (muscles and tendons). Stretching exercise for all muscles was repeated ten times during session.
3. Passive range of motion: The wrist and fingers were moved slowly, gently and smoothly in all directions passively through the available range of motion. Passive range of motion was applied for five minutes at beginning and for five minutes at the end of session.
4. Active range of motion: Patient was asked to perform wrist flexion, extension, radial and ulnar deviation as well as fingers flexion, extension and abduction actively as much as possible for two sets each set ten repetitions (i.e. twenty repetitions at beginning of session and twenty repetitions at end of session).
5. Edema control: hand was elevated on towel with pressure applied to the volar and dorsum of the hand with passive ROM applied by the examiner firstly then patients was asked to perform flexion and extension of fingers for fifteen repetitions of fifteen second relax for three times.

Group II received Russian current stimulation in addition to traditional exercise:

Electrical stimulation was carried out using phyaction 787 device (Manufactured by Uniphy, serial number 24823, Netherlands). Two equal sized carbon rubber electrodes were placed on common flexor origin (below medial epicondyle of humerus) and the other on distal part of flexor carpi radialis and flexor carpi ulnaris, perpendicular to the longitudinal axis of the forearm for fifteen minutes time of stimulation. The frequency was 2.5 kHz, with a burst duty cycle of 50% and intensity adjusted according to patient tolerant. The burst duration is 10 milliseconds at 50 Hz.

Group III received closed kinetic chain exercise plus traditional exercise:

1. Wall press exercise: The patient stood with feet shoulder-width apart, arms held directly out in front of the body at 90º of elevation against the wall. Feet are approximately two to three feet (0.6-0.9 meter) away from the wall. The patient pressed on the wall with the distal extremity fixed on stable surface and asked to keep pressing for thirty seconds.
2. Plyometric wall push-up exercise: The patient stood away from the wall by about two feet with both arms in front of body at approximately 90o. The chest was lowered toward the wall until the elbows were bent approximately 45º to 60º. The patient then forcefully pushed the wall to return to starting position.
3. Quadruped rhythmic stabilization exercise: Patient on hands and knees on a table or floor with the head and spine kept in neutral position. The examiner instruct the patient to hold the body without any movement. Against short, rapid pushing motions from side to side, front to back, and along diagonals. The pushing motions progressed from submaximal to maximal intensities and from slow to fast. The patient was asked to preserve the balance while the exercise maintained for thirty seconds, and each week the time increased by five seconds for progression.
4. Push up exercise: Quadruped on a plinth or on the floor. The patient lowered the body into arms until the elbows bent approximately 45º to 60º. The patient then pushed the floor to return to the starting position.

All patients in the three groups were applied the program 3 timed a weak.

CKC exercises performed ten times and each week two more repetitions added as a progression.

The aim of this study was explained and informed consent was obtained from all patients.

Outcome Measures Pain, functional disability, ROM measurements (wrist flexion-extension, radial-ulnar deviation), and grip strength of injured hand were used as outcome measures. Pre-treatment (baseline) and post- treatment (after six weeks) measurements were recorded.

Pain and functional disability Patient rated wrist evaluation (PRWE) questionnaire: The PRWE questionnaire considered a subjective outcome measure consisting of fifteen questions answered on a scale of one to ten. Five questions focus on wrist pain, and ten questions focus on function. The patient was asked to describe the pain as well as the function of the involved hand on the scale and the answered numbers for pain and function were calculated for each one separately for analysis.

Range of Motion Baseline digital goniometer (Baseline ®, Aurora, IL, USA) for assessment of wrist ROM; flexion, extension [14], radial and ulnar deviation [15]. The device displays 0 to 180 degrees on an LCD screen for viewing readings, and has the ability to freeze angle measurements for reference. The goniometer has a durable powder-coated steel or plastic exterior with inch/cm marks screened on its arms.

Grip Strength A Jamar dynamometer for measurement of grip strength in kilograms (Jamar, J.A. Preston Co., Michigan, USA) [16,17]. The maximal muscle strength was measured with elbow flexion 90°, and wrist placed in neutral position [18].

Range of motion and grip strength performed for 3 repetitions and the mean of the three trials was record.

ELIGIBILITY:
Inclusion Criteria:

* patients with stable colles' fractures treated conservatively with closed reduction

Exclusion Criteria:

1. Patient less than 20 years old.
2. Intraarticular fracture of involved hand.
3. Any problem affects shoulder /elbow joints of the involved side.
4. Nerve lesions.
5. Fracture of the ulna.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Patient rated wrist evaluation (PRWE) questionnaire | 6 weeks

SECONDARY OUTCOMES:
Baseline digital goniometer (Baseline ®, Aurora, IL, USA) for assessment of wrist ROM | 6 weeks

OTHER OUTCOMES:
A Jamar dynamometer for measurement of grip strength in kilograms | 6 weeks

REFERENCES:
- [Background] Belloti JC, Santos JB, Atallah AN, Albertoni WM, Faloppa F. Fractures of the distal radius (Colles' fracture). Sao Paulo Med J. 2007 May 3;125(3):132-8. doi: 10.1590/s1516-31802007000300002. PMID 17923936